CLINICAL TRIAL: NCT01622699
Title: Implementation of a Transcutaneous Bilirubinometer in Jaundiced Newborns: a Randomised Controlled Trial
Brief Title: Implementation of a Transcutaneous Bilirubinometer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Amalia Children's Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: TcB AmaliaCC
Record Dates: First submitted 2012-06-12; First posted 2012-06-19 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Neonatal Jaundice; Hyperbilirubinemia
Keywords: Jaundice; Neonatal Jaundice; Hyperbilirubinemia; Transcutaneous bilirubin measurement; Transcutaneous bilirubinometry; jaundice meter; Visual assessment of bilirubin; Newborn
MeSH Terms: conditions — Jaundice, Neonatal; Hyperbilirubinemia; Jaundice

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcutaneous bilirubin measurements (Experimental): In this intervention group, the initial visual assessment of jaundice wille be followed by measurement by transcutaneous bilirubinometer
  Interventions: Device: Transcutaneous Bilirubinometer
- Visual assessment of neonatal jaundice (Active Comparator): In this control group (standard of care) the visual assessment will be followed by measurement of blood bilirubin as indicated by the physician
  Interventions: Other: visual assessment of neonatal jaundice

INTERVENTIONS:
Device: Transcutaneous Bilirubinometer — If a baby is jaundiced, the ward-nurse will perform a transcutaneous bilirubin measurement. It takes about 5 seconds to perform the measurement at the forehead or sternum of the baby. The device is a validated measurement-tool, which provides us with an estimated serum bilirubin-concentration. This is not an invasive procedure: A light-reflection is used to measure transcutaneous bilirubin.
  Other Names: JaundiceMeter-103®, Dräger
  Arms: Transcutaneous bilirubin measurements
Other: visual assessment of neonatal jaundice — To detect newborns with jaundice (who will possibly meet the criteria for phototherapy) there have been international guidelines formulated by the American Academy of Pediatrics. The standard of care at the neonatal- and maternity ward of our hospital to detect those newborns is visual assessment according to these guidelines.
  Arms: Visual assessment of neonatal jaundice

SUMMARY:
Neonatal jaundice, caused by hyperbilirubinemia, is frequently seen in healthy newborns. Assessment of the degree of jaundice is usually done visually,and if necessary serum bilirubin is investigated in a blood sample. The visual assessment is subjective and can alternatively be replaced by transcutaneous measurement.The transcutaneous bilirubinometer is a validated measurement-tool, which provides us with an estimated serum bilirubin-concentration. Little is known about the effect of the actual use of a bilirubinometer on the quality of care. Further evidence is needed to evaluate whether transcutaneous bilirubin measurements improve clinical outcome (use of blood tests, phototherapy and exchange transfusion), shorten length of stay and reduce costs. Therefore we aim to perform a Randomized controlled trial to evaluate the cost-effectiveness of implementing the use of a transcutaneous bilirubinometer in jaundiced neonates, a gestational age of 32 weeks. The assessment of jaundice by use of a transcutaneous bilirubinometer is compared to visual assessment of jaundice

DETAILED DESCRIPTION:
Rationale:

Neonatal jaundice, caused by hyperbilirubinemia, is frequently seen in healthy newborns. Severe hyperbilirubinemia can cause bilirubin encephalopathy (kernicterus). Assessment of the degree of jaundice is usually done visually,and if necessary serum bilirubin is investigated in a blood sample. The visual assessment is subjective and can alternatively be replaced by transcutaneous measurement.The transcutaneous bilirubinometer is a validated measurement-tool, which provides us with an estimated serum bilirubin-concentration. Little is known about the effect of the actual use of a bilirubinometer on the quality of care. Further evidence is needed to evaluate whether transcutaneous bilirubin measurements improve clinical outcome (use of blood tests, phototherapy and exchange transfusion), shorten length of stay and reduce costs.

Objective:

To evaluate the cost-effectiveness of implementing the use of a transcutaneous bilirubinometer in jaundiced neonates.

Study design:

Randomized controlled trial

Study population:

All jaundiced newborns beyond a gestational age of 32 weeks and younger than 8 days who are admitted at the maternity-ward or the neonatal-ward of our hospital.

Intervention:

Assessment of jaundice by use of a transcutaneous bilirubinometer.

Control:

Visual assessment of jaundice (current standard of care)

Main study parameters/endpoints:

Primary outcome variable:

The number of blood punctures for bilirubin measurement.

Secondary outcome:

Phototherapy duration in hours, amount of bilirubin-values above the exchange transfusion limit, highest measured serum bilirubin, costs (blood test, use bilirubinometer, costs admittance)

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Burden: A non-invasive transcutaneous measurement using a transcutaneous bilirubinometer (harmless light-reflection-technique). It takes at most 5 seconds to perform the measurement at the forehead or sternum.

Risk:It could be possible that a severe hyperbilirubinemia will be missed. This is a greater risk in the control group, due to the fact that visual assessment is known to be unreliable. When in doubt, the clinical team will have the authority to determine the serum bilirubin-value.

ELIGIBILITY:
Inclusion Criteria:

* All newborns at the pediatric- and maternity-ward with visible jaundice.
* Gestational age of 32 weeks or more.
* Older than 24 hours.
* Younger than 8 days.

Exclusion Criteria:

* Neonatal jaundice within 24 hours or after 8 days
* Hemolysis present based on maternal history (for example irregular erythrocyte antibodies)
* Bilirubin encephalopathy
* Newborns during/after phototherapy
* Large congenital anomaly at forehead/sternum
* Serum bilirubin-value is already known before admission to the pediatric ward;those newborns are to be admitted because the serum bilirubin-level has reached the phototherapy or exchange transfusion limit.

Ages: 24 Hours to 8 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 430 (Actual)
Dates: Start 2013-10; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jolita Bekhof, MD, Principal Investigator — Isala
Locations (1):
- Isala Klinieken, Amalia Childrens Clinic, Zwolle, Overijssel, Netherlands

REFERENCES:
- [Background] American Academy of Pediatrics Subcommittee on Hyperbilirubinemia. Management of hyperbilirubinemia in the newborn infant 35 or more weeks of gestation. Pediatrics. 2004 Jul;114(1):297-316. doi: 10.1542/peds.114.1.297. PMID 15231951
- [Background] Dijk PH, de Vries TW, de Beer JJ; Dutch Pediatric Association. [Guideline 'Prevention, diagnosis and treatment of hyperbilirubinemia in the neonate with a gestational age of 35 or more weeks']. Ned Tijdschr Geneeskd. 2009;153:A93. Dutch. PMID 19785881
- [Background] Szabo P, Wolf M, Bucher HU, Fauchere JC, Haensse D, Arlettaz R. Detection of hyperbilirubinaemia in jaundiced full-term neonates by eye or by bilirubinometer? Eur J Pediatr. 2004 Dec;163(12):722-7. doi: 10.1007/s00431-004-1533-7. PMID 15365826
- [Derived] van den Esker-Jonker B, den Boer L, Pepping RM, Bekhof J. Transcutaneous Bilirubinometry in Jaundiced Neonates: A Randomized Controlled Trial. Pediatrics. 2016 Dec;138(6):e20162414. doi: 10.1542/peds.2016-2414. Epub 2016 Nov 4. PMID 27940715

RESULTS

PARTICIPANT FLOW:
Groups:
- Transcutaneous Bilirubin Measurements: patients that were randomized to get bilirubinemeasurements through the transcutaneous bilirubinometer
- Visual Assessment of Neonatal Jaundice: pateients that were randomized to the standrad treatemnt, thus withoutthe use of the transcutaneous bilirubinometer
Period: Overall Study
Arm/Group | Transcutaneous Bilirubin Measurements | Visual Assessment of Neonatal Jaundice
Started | 213 | 217
Completed | 213 | 217
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Transcutaneous Bilirubin Measurements: patients that were randomized to get bilirubine measurements through the transcutaneous bilirubinometer
- Visual Assessment of Neonatal Jaundice: patients that were randomized NOT to get bilirubinemeasurements through the transcutaneous bilirubinometer
- Total: Total of all reporting groups
Arm/Group | Transcutaneous Bilirubin Measurements | Visual Assessment of Neonatal Jaundice | Total
Number analyzed (Participants) | 213 | 217 | 430
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 213 | 217 | 430
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: hours] — age at first measurement of bilirubin (either through bloodpuncture or transcutaneous bilirubinometer)
  hours
    agee | 53.9 (17.4) | 59.2 (19.8) | 56.6 (18.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 98 | 201
  Male | 110 | 119 | 229
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 213 | 217 | 430

OUTCOME MEASURES:

1. Primary Outcome: Number of Blood Tests for Bilirubin Measurement (Before the Potential Start of Phototherapy).
Time Frame: up to 1 year
Measure: Median (Inter-Quartile Range); unit: blood tests for bilirubin
Arm/Group | Transcutaneous Bilirubin Measurements | Visual Assessment of Neonatal Jaundice
Number analyzed (Participants) | 213 | 217
blood tests for bilirubin | 0 [0 to 2] | 1 [1 to 2]

2. Secondary Outcome: Number of Patients With Serum Bilirubin-values Above the 'Exchange Transfusion Limit'
Time Frame: up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Transcutaneous Bilirubin Measurements | Visual Assessment of Neonatal Jaundice
Number analyzed (Participants) | 213 | 217
Participants | 3 | 1

3. Secondary Outcome: Highest Measured Serum Bilirubin-value
Time Frame: up to 1 year
Measure: Mean (Standard Deviation); unit: micromol/l
Arm/Group | Transcutaneous Bilirubin Measurements | Visual Assessment of Neonatal Jaundice
Number analyzed (Participants) | 213 | 217
micromol/l | 210 (46) | 217 (65)

4. Secondary Outcome: Number of Patients Having Kernicterus
Description: Kernicterus is a very rare condition. As it is a possible complication of neonatal hyperbilirubinemia, it's an outcome measure.
Time Frame: up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Transcutaneous Bilirubin Measurements | Visual Assessment of Neonatal Jaundice
Number analyzed (Participants) | 213 | 217
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 weeks
Groups:
- Transcutaneous Measurement: patients that were randomized to get bilirubinemeasurements through the transcutaneous bilirubinometer
Arm/Group | Transcutaneous Measurement | Visual Assessment of Neonatal Jaundice
All-Cause Mortality (participants affected / at risk) | 0/213 | 0/217
Serious Adverse Events (participants affected / at risk) | 0/213 | 0/217
Other Adverse Events (participants affected / at risk) | 0/213 | 0/217

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes